CLINICAL TRIAL: NCT06824012
Title: Development and Evaluation of a Daily-Activity-Based Growth Mindset Intervention for Adolescents and Staff in Youth Custody Frameworks: A Mixed-Methods Study
Brief Title: Development and Evaluation of a Growth Mindset Intervention for Adolescents in Youth Custody Frameworks: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miri Tal-Saban (Other)
Responsible Party: Sponsor-Investigator, Miri Tal-Saban, Principal Investigator, Hebrew University of Jerusalem
Organization: Hebrew University of Jerusalem (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5032023
Record Dates: First submitted 2025-02-11; First posted 2025-02-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: At Risk Youth
Keywords: Growth Mindset; Adolescent Behavior; Youth in Custody; Psychological Adaptation; Daily Activities; Resilience
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Growth Mindset Intervention Group (Experimental): Participants in this arm will receive a structured, daily-activity-based intervention designed to promote a growth mindset. The intervention includes:
  Guided participation in meaningful daily activities tailored to individual needs.
  Reflective discussions and feedback sessions to reinforce growth mindset principles.
  Pre- and post-intervention assessments using the Canadian Occupational Performance Measure (COPM) and structured questionnaires. The aim is to enhance psychological adaptation, resilience, and daily life participation among adolescents in youth custody frameworks and their staff.
  Interventions: Behavioral: Growth Mindset Intervention

INTERVENTIONS:
Behavioral: Growth Mindset Intervention — A structured, daily-activity-based intervention program designed to foster a growth mindset among adolescents in youth custody frameworks and their staff. The intervention involves:
  Guided engagement in practical, meaningful daily activities tailored to individual and group needs.
  Reflective feedback sessions to reinforce principles of a growth mindset. Pre- and post-intervention assessments using standardized tools, including the Canadian Occupational Performance Measure (COPM) and structured questionnaires.

SUMMARY:
The purpose of this study is to develop and evaluate a daily-activity-based intervention aimed at fostering a growth mindset among adolescents in youth custody frameworks and their staff. The study seeks to answer whether this intervention can improve participants' perceptions of their ability to adapt, enhance daily life participation, and identify barriers and facilitators for promoting a growth mindset in this unique population. Using a mixed-methods design, the study includes pre- and post-intervention assessments with the Canadian Occupational Performance Measure (COPM), structured questionnaires, and focus groups to evaluate the effectiveness of the program.

DETAILED DESCRIPTION:
This study aims to develop and evaluate an intervention program designed to promote a growth mindset among adolescents residing in youth custody frameworks and their staff. The intervention is grounded in daily-activity-based approaches, emphasizing practical engagement in meaningful activities and reflective learning. The program is tailored to address the unique challenges and strengths of participants within these frameworks, with the goal of fostering adaptability, resilience, and improved participation in daily life tasks.

The research employs a mixed-methods design to comprehensively assess the intervention's impact. Quantitative data will be collected using the Canadian Occupational Performance Measure (COPM) to measure changes in participants' perceptions of their performance and satisfaction with daily tasks. Structured pre- and post-intervention questionnaires will further evaluate shifts in growth mindset attitudes. Qualitative data will be gathered through focus groups with adolescents, alumni, and staff, providing insights into the intervention's feasibility, perceived barriers, and opportunities for adaptation.

The study is conducted at two youth custody institutions, Alma and Mitspa-Yam, which provide residential care for adolescents in high-risk situations. Participants include adolescents currently in care, alumni, and staff members. Findings from this research are expected to inform the development of evidence-based guidelines for integrating growth mindset interventions into youth custody settings, with implications for enhancing long-term outcomes for participants.

ELIGIBILITY:
Inclusion Criteria:

Adolescents currently residing in youth custody frameworks who are selected by the institution's staff based on their suitability for the study.

Alumni of youth custody frameworks who are contacted directly by the research team.

Exclusion Criteria:

Adolescents whose mental or physical condition prevents them from participating in the study.

Individuals who are unable to complete questionnaires or reflectively describe their experiences.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM). | Before and after the intervention (approximately 8 weeks).
  This measure evaluates changes in participants' perceptions of their daily task performance and satisfaction before and after the intervention.
  Scale Details:
  Scale Title: COPM Performance and Satisfaction Scales Range: 1 to 10 Interpretation: Higher scores indicate better performance and greater satisfaction.
  Time Frame: Before and after the intervention (approximately 8 weeks).

SECONDARY OUTCOMES:
Analysis of Barriers and Facilitators in the Framework - Customized Survey Scale | Before and after the intervention (approximately 8 weeks).
  his measure assesses perceived barriers and facilitators in the context of daily activities, psychological adaptation, and interpersonal support within the youth custody framework. The survey evaluates aspects such as perceived trust in staff, sense of security, support from peers and staff, independence, organization, and expectations for the future.
  Scale Details:
  Scale Title: Youth Custody Resident Experience Survey (YCRES) Range: 1 (Strongly Disagree) to 10 (Strongly Agree) Interpretation: Higher scores indicate a more positive perception of facilitators (e.g., trust in staff, support from peers, self-efficacy), whereas lower scores suggest greater perceived barriers and difficulties in adaptation.

CONTACTS AND LOCATIONS:
Locations (1):
- Alma Boarding School, Ashdod, Israel, Israel

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns related to the sensitive nature of the data collected from adolescents in youth custody frameworks. Additionally, restrictions imposed by the ethics committee and institutional guidelines prevent the sharing of such data.

REFERENCES:
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506
- [Background] Burnette JL, O'Boyle EH, VanEpps EM, Pollack JM, Finkel EJ. Mind-sets matter: a meta-analytic review of implicit theories and self-regulation. Psychol Bull. 2013 May;139(3):655-701. doi: 10.1037/a0029531. Epub 2012 Aug 6. PMID 22866678
- [Background] Bowman J, Mogensen L, Marsland E, Lannin N. The development, content validity and inter-rater reliability of the SMART-Goal Evaluation Method: A standardised method for evaluating clinical goals. Aust Occup Ther J. 2015 Dec;62(6):420-7. doi: 10.1111/1440-1630.12218. Epub 2015 Aug 19. PMID 26286379
- [Background] Billingsley, J., Lipsey, N. P., Burnette, J. L., & Pollack, J. M. (2021). Growth mindsets: defining, assessing, and exploring effects on motivation for entrepreneurs and nonentrepreneurs. Current Psychology, 42(11), 8855-8873. https://doi.org/10.1007/s12144-021-02149-w